CLINICAL TRIAL: NCT04728529
Title: Septic Shock Management Guided by Ultrasound: A Randomized Control Trial (SEPTICUS Trial)
Brief Title: Septic Shock Management Guided by Ultrasound: SEPTICUS Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saptadi Yuliarto (Other)
Responsible Party: Sponsor-Investigator, Saptadi Yuliarto, Head of Pediatric Emergency and Intensive Care Department, University of Brawijaya
Organization: University of Brawijaya (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University of Brawijaya
Record Dates: First submitted 2020-12-31; First posted 2021-01-28 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Septic Shock
Keywords: septic shock; Doppler ultrasonography; Fluid resuscitation; Vasoactive therapy; Mortality rate; Fluid overload
MeSH Terms: conditions — Shock, Septic; Edema

STUDY DESIGN:
Intervention Model Description: Each eligible patient will be randomized into 2 groups of treatment, the USSM protocol or the ACCM protocol. All of subjects in each group will receive emergency management: oxygen support, vascular access, and fluid resuscitation. In intervention group, each step of fluid and vasoactive management will be guided by clinical sign and Doppler ultrasonography, whereas in control group only guided by the clinical sign.
Masking Description: Outcome of mortality rate, macrocirculation hemodynamic parameter, and microcirculation laboratory parameter are objective measurement (does not influenced by assessors's subjectiveness).
  However, the assessor of liver enlargement and lung US score will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- USSM protocol (Experimental): patient in the intervention group receive fluid resuscitation and inotropic-vasoactive agent, if needed, in accordance to USSM protocol of fluid resuscitation.
  Interventions: Procedure: USSM protocol
- ACCM protocol (Experimental): patient in the control group receive fluid resuscitation and inotropic-vasoactive agent, if needed, in accordance to ACCM protocol of fluid resuscitation.
  Interventions: Procedure: ACCM protocol

INTERVENTIONS:
Procedure: USSM protocol — In the initial step, all subjects will receive emergency management: oxygen support, vascular access, and fluid therapy. Doppler ultrasonography by Ultrasound Cardiac Output Monitoring (USCOM) is also performed to record initial stroke volume (SV), cardiac index (CI), and systemic vascular resistance (SVR). The initial fluid resuscitation is 20 mL/kg body weight, then the response measured by clinical and USCOM examination. If any improvement of clinical sign and normal SVI, CI, SVR, intervention will be stopped. In contrary, if shock persist, subsequent fluid resuscitation and/or vasoactive therapy will be administered, guided by USCOM.
  The therapeutic goal of USCOM: SVI 30-60 mL/m2, CI 3.3-6.0 L/minute/m2, and SVRI 800-1600 d.s/cm5/m2
  Arms: USSM protocol
Procedure: ACCM protocol — In the initial step, all subjects will receive emergency management: oxygen support, vascular access, and fluid therapy. Doppler ultrasonography by Ultrasound Cardiac Output Monitoring (USCOM) is also performed to record initial stroke volume (SV), cardiac index (CI), and systemic vascular resistance (SVR). The initial fluid resuscitation is 20 mL/kg body weight, then the response measured by clinical. If any improvement of clinical sign, intervention will be stopped. In contrary, if shock persist, subsequent fluid resuscitation and/or vasoactive therapy will be administered, guided by clinical parameter.
  Arms: ACCM protocol

SUMMARY:
This clinical study aims to compare the recent septic shock management protocol from American College of Critical Care Medicine (ACCM) to Ultrasound-guided Septic Shock Management (USSM) protocol. USSM protocol laid on Doppler ultrasonography to evaluate stroke volume, cardiac index, and systemic vascular resistance in each step of management to decide the proper fluid resuscitation and vasoactive therapy; differs from ACCM protocol which use clinical finding in its early step. ACCM protocol application elicits risk of improper therapy since clinical sign per se often could not describe the certain cardiac output. This can be prevented earlier by USSM protocol. The outcome compared of the two protocols is: mortality rate, clinical parameter, macrocirculation hemodynamic parameter, laboratory microcirculation parameter, and signs of fluid overload. The investigators hypothesized if the USSM protocol had a better outcome and less fluid overload complication.

DETAILED DESCRIPTION:
This study is a randomized controlled trial to compare the usage of ACCM protocol and USSM protocol in fluid resuscitation for septic shock pediatric patients. The USSM protocol is the intervention, and the ACCM protocol is the control. This study implemented in septic shock pediatric patients treated in the intensive care unit. Each patient will be randomized into 2 groups, the USSM group or the ACCM group. In the initial step, all patient in each group will receive early acute/emergency therapy: oxygen support, vascular access, and fluid resuscitation. The monitoring of the patient including clinical parameters and laboratory examination for both groups, except Doppler ultrasonography that performed in each step of management of the intervention group. The monitoring is performed every 15 minutes in the first hour of resuscitation. If the patient show good response (fluid responsive shock), the monitoring stops in 1 hour. In contrast, if the patient reveal fluid refractory shock, the vasoactive agent will be administered and monitoring continues until 6 hours. All outcome parameters, except mortality rate, will be recorded at 6 hours. The mortality rates will be recorded at 72 hours and time of intensive care discharge.

Sample size in this study was calculated by clinical trial formula for mortality rate with a significance level of 0.05 and study power of 0.2. From the calculation, the subject needed is 170 patients for each group (total 340 subjects). The basic characteristics of the patient will be analyzed descriptively. All parameter data will be analyzed statistically by Statistical Product and Service Solution (SPSS) 20, preceded by normality test and homogeneity test. The study analysis will be intention-to-treat. The mortality rate was analyzed by Kaplan-Meier survival analysis. Data transformation will be performed if needed in case of outlier data or out-of-range results.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as septic shock according to Pediatric Surviving Campaign (2005)

Exclusion Criteria:

* patient with uncorrected congenital heart disease with shunting
* obtain fluid resuscitation before recruitment process
* obtain inotropic-vasoactive agent before recruitment process
* after undergo any heart surgery

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 72 hours of the initial fluid resuscitation
  Time of mortality occurrence since randomization, comparing intervention and control group.
Number of mortality | 72 hours of the initial fluid resuscitation
  Amount of non-survivor subject, comparing intervention and control group.

SECONDARY OUTCOMES:
Heart rate | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Heart rate is measured by vital sign monitor device, reported in beat/minute, and classified into bradycardia (below normal rate according to age of PALS criteria), normal, and tachycardia (above normal rate according to age of PALS criteria).
Capillary refill time | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Capillary refill time is measured by pressing forehead and sternal skin; time needed for the pink color to return will be measured and reported in second, then classified based on WHO criteria, into prolonged (above 3 seconds) or normal (below or equal than 3 seconds).
Peripheral pulse strength | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Peripheral pulse strength is measured by comparing peripheral radial pulse and central (carotid or femoral) pulse, reported qualitatively as weak or normal/strong
Systolic blood pressure | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Systolic blood pressure is measured by vital sign monitor device and reported in mmHg, and classified into hypotension (below 5th percentiles according to age of PALS criteria), normal (above or equal than 5th percentiles according to age of PALS criteria), and high (above 95th percentiles according to age of PALS criteria).
Mean arterial pressure | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Mean arterial pressure (MAP) is measured by vital sign monitor device and reported in mmHg, and classified into hypotension (below 5th percentiles according to age of PALS criteria), normal (above or equal than 5th percentiles according to age of PALS criteria), and high (above 95th percentiles according to age of PALS criteria).
Systemic vascular resistance index | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Systemic vascular resistance index (SVRI) is measured by USCOM, reported in d.s/cm5/m2, and classified into low (below 800), normal (800 to 1600), and high (above 1600)
Stroke volume index | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Stroke volume index (SVI) is measured by USCOM, reported in mL/m2, and classified into low (below 30), normal (30 to 60), and high (above 60).
Cardiac index | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Cardiac index (CI) is measured by USCOM, reported in L/minute/m2, and classified into low (below 3.3), normal (3.3 to 6.0), and high (above 6.0).
Base deficit | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Base deficit is measured by blood gas analysis examination, reported in mmol/L, and classified into low (below -3), normal (-3 to 3), and high (above 3).
Blood lactate level | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Blood lactate level is measured from arterial blood, reported in mmol/L, and classified into normal (below or equal to 2.0) or high (above 2.0).
Liver span increase | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  The increase of liver span is clinically measured from mid-costal right arch to the edge of liver, and reported in centimeters.
Lung ultrasound score | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  Lung Ultrasound Score is examined with ultrasound using linear transducer (7.5 to 11 Mhz) to measure pulmonary parenchyma aeration on 12 scan areas (6 areas in each hemithorax), by a doctor who is ultrasound-certified lung. Each hemithorax is divided by 3 vertical lines (parasternal, anterior axillary, and posterior axillary) so that it becomes 3 areas (anterior, lateral, and posterior); and 1 horizontal line dividing the hemithorax into 2 equal parts. In each area a score is recorded. The final result is a total score of 12 areas. The scores are stated as follows:
  i. 0 = no (or very few) B-lines ii. 1 = B-lines look many but separate (separated B-lines) iii. 2 = many B-lines and converge (coalescent B-lines) iv. 3 = lung consolidation
Vasoactive-inotropic score (VIS) | 1 hour in fluid-responsive subject or 6 hour in fluid-refractory subject after fluid resuscitation initiated
  The Vasoactive-Inotropic Score (VIS), quantifies the amount of cardiovascular support required by subjects and includes dopamine, dobutamine, epinephrine, milrinone, vasopressin, and norepinephrine.

CONTACTS AND LOCATIONS:
Overall Officials: Saptadi Yuliarto, MD, Study Director — University of Brawijaya
Locations (1):
- RSUD dr. Saiful Anwar, Malang, East Java, Indonesia

REFERENCES:
- [Background] Davis AL, Carcillo JA, Aneja RK, Deymann AJ, Lin JC, Nguyen TC, Okhuysen-Cawley RS, Relvas MS, Rozenfeld RA, Skippen PW, Stojadinovic BJ, Williams EA, Yeh TS, Balamuth F, Brierley J, de Caen AR, Cheifetz IM, Choong K, Conway E Jr, Cornell T, Doctor A, Dugas MA, Feldman JD, Fitzgerald JC, Flori HR, Fortenberry JD, Graciano AL, Greenwald BM, Hall MW, Han YY, Hernan LJ, Irazuzta JE, Iselin E, van der Jagt EW, Jeffries HE, Kache S, Katyal C, Kissoon N, Kon AA, Kutko MC, MacLaren G, Maul T, Mehta R, Odetola F, Parbuoni K, Paul R, Peters MJ, Ranjit S, Reuter-Rice KE, Schnitzler EJ, Scott HF, Torres A Jr, Weingarten-Arams J, Weiss SL, Zimmerman JJ, Zuckerberg AL. American College of Critical Care Medicine Clinical Practice Parameters for Hemodynamic Support of Pediatric and Neonatal Septic Shock. Crit Care Med. 2017 Jun;45(6):1061-1093. doi: 10.1097/CCM.0000000000002425. PMID 28509730
- [Background] Weiss SL, Peters MJ, Alhazzani W, Agus MSD, Flori HR, Inwald DP, Nadel S, Schlapbach LJ, Tasker RC, Argent AC, Brierley J, Carcillo J, Carrol ED, Carroll CL, Cheifetz IM, Choong K, Cies JJ, Cruz AT, De Luca D, Deep A, Faust SN, De Oliveira CF, Hall MW, Ishimine P, Javouhey E, Joosten KFM, Joshi P, Karam O, Kneyber MCJ, Lemson J, MacLaren G, Mehta NM, Moller MH, Newth CJL, Nguyen TC, Nishisaki A, Nunnally ME, Parker MM, Paul RM, Randolph AG, Ranjit S, Romer LH, Scott HF, Tume LN, Verger JT, Williams EA, Wolf J, Wong HR, Zimmerman JJ, Kissoon N, Tissieres P. Surviving Sepsis Campaign International Guidelines for the Management of Septic Shock and Sepsis-Associated Organ Dysfunction in Children. Pediatr Crit Care Med. 2020 Feb;21(2):e52-e106. doi: 10.1097/PCC.0000000000002198. PMID 32032273
- [Background] Weiss SL, Peters MJ, Alhazzani W, Agus MSD, Flori HR, Inwald DP, Nadel S, Schlapbach LJ, Tasker RC, Argent AC, Brierley J, Carcillo J, Carrol ED, Carroll CL, Cheifetz IM, Choong K, Cies JJ, Cruz AT, De Luca D, Deep A, Faust SN, De Oliveira CF, Hall MW, Ishimine P, Javouhey E, Joosten KFM, Joshi P, Karam O, Kneyber MCJ, Lemson J, MacLaren G, Mehta NM, Moller MH, Newth CJL, Nguyen TC, Nishisaki A, Nunnally ME, Parker MM, Paul RM, Randolph AG, Ranjit S, Romer LH, Scott HF, Tume LN, Verger JT, Williams EA, Wolf J, Wong HR, Zimmerman JJ, Kissoon N, Tissieres P. Surviving sepsis campaign international guidelines for the management of septic shock and sepsis-associated organ dysfunction in children. Intensive Care Med. 2020 Feb;46(Suppl 1):10-67. doi: 10.1007/s00134-019-05878-6. PMID 32030529
- [Background] Santhanam I, Sangareddi S, Venkataraman S, Kissoon N, Thiruvengadamudayan V, Kasthuri RK. A prospective randomized controlled study of two fluid regimens in the initial management of septic shock in the emergency department. Pediatr Emerg Care. 2008 Oct;24(10):647-55. doi: 10.1097/PEC.0b013e31818844cf. PMID 19242131
- [Background] Ranjit S, Aram G, Kissoon N, Ali MK, Natraj R, Shresti S, Jayakumar I, Gandhi D. Multimodal monitoring for hemodynamic categorization and management of pediatric septic shock: a pilot observational study*. Pediatr Crit Care Med. 2014 Jan;15(1):e17-26. doi: 10.1097/PCC.0b013e3182a5589c. PMID 24196006
- [Background] Ceneviva G, Paschall JA, Maffei F, Carcillo JA. Hemodynamic support in fluid-refractory pediatric septic shock. Pediatrics. 1998 Aug;102(2):e19. doi: 10.1542/peds.102.2.e19. PMID 9685464
- [Background] Horster S, Stemmler HJ, Strecker N, Brettner F, Hausmann A, Cnossen J, Parhofer KG, Nickel T, Geiger S. Cardiac Output Measurements in Septic Patients: Comparing the Accuracy of USCOM to PiCCO. Crit Care Res Pract. 2012;2012:270631. doi: 10.1155/2012/270631. Epub 2011 Nov 29. PMID 22191019
- [Background] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT04728529/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT04728529/ICF_000.pdf